CLINICAL TRIAL: NCT05670509
Title: Intranasal vs Buccal vs Intramuscular Midazolam for the Home and Emergency Treatment of Acute Seizures in Pediatric Egyptian Patients
Brief Title: Intranasal vs Buccal vs Intramuscular Midazolam for the Home and Emergency Treatment of Acute Seizures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fmasu md 19 1 2019
Record Dates: First submitted 2022-10-08; First posted 2023-01-04 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2022-12

CONDITIONS: Convulsions
MeSH Terms: conditions — Seizures | interventions — Group Homes

STUDY DESIGN:
Intervention Model Description: Two major groups were included (home and ER group) and each were subdivided into 3 groups according to route of administration (nasal, buccal and IM)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Nasal administration of midazolam in home group (Experimental): treatment with intranasal midazolam in children with known seizure disorder who were prescribed midazolam by pediatric neurologist at home with doses of 0.2 mg/kg (maximum, 10 mg) body weight of the standard IV formulation of midazolam (5mg/mL) via a metered dose sprayer at 0.1 mL/spray (i.e. 0.5mg/spray). If the volume to be administered exceeded 1 mL, then the dose was divided between both nostrils to avoid runoff and swallowing. children with known seizure disorder who were prescribed midazolam by pediatric neurologist
  Interventions: Drug: administration of Nasal midazolam in home group as a rescue medication for seizure control.
- buccal administration of midazolam in home group (Experimental): treatment with buccal midazolam in children with known seizure disorder who were prescribed midazolam by pediatric neurologist at home with doses of 0.2 mg/kg (maximum, 10 mg) body weight of the standard IV formulation of midazolam (5mg/mL) via dripping between the cheek and the gum per side using insulin syringe
  Interventions: Drug: administration of Buccal midazolam in home group as a rescue medication for seizure control.
- intramuscular administration of midazolam in home group (Experimental): treatment with intramuscular midazolam in children with known seizure disorder who were prescribed midazolam by pediatric neurologist at home with doses of 0.2 mg/kg (maximum, 10 mg) body weight of the standard IV formulation of midazolam (5mg/mL) administered via using 3 mm syringe in the front aspect of thigh
  Interventions: Drug: administration of intramuscular midazolam in homegroup as a rescue medication for seizure control.
- Nasal administration of midazolam in ER group (Experimental): treatment with intranasal midazolam in children presenting to ER with acute seizures with doses of 0.2 mg/kg (maximum, 10 mg) body weight of the standard IV formulation of midazolam (5mg/mL) via a metered dose sprayer at 0.1 mL/spray (i.e. 0.5mg/spray). If the volume to be administered exceeded 1 mL, then the dose was divided between both nostrils to avoid runoff and swallowing.
  Interventions: Drug: administration of Nasal midazolam in ER group as a rescue medication for seizure control.
- buccal administration of midazolam in ER group (Experimental): treatment with buccal midazolam in children presenting to ER with acute seizures with doses of 0.2 mg/kg (maximum, 10 mg) body weight of the standard IV formulation of midazolam (5mg/mL) via dripping between the cheek and the gum per side using insulin syringe
  Interventions: Drug: administration of Buccal midazolam in ER group as a rescue medication for seizure control.
- Intramuscular administration of midazolam in ER group (Experimental): treatment with intramuscular midazolam in children presenting to ER with acute seizures with doses of 0.2 mg/kg (maximum, 10 mg) body weight of the standard IV formulation of midazolam (5mg/mL) administered via using 3 mm syringe in the front aspect of thigh
  Interventions: Drug: administration of intramuscular midazolam in ER group as a rescue medication for seizure control.

INTERVENTIONS:
Drug: administration of Nasal midazolam in home group as a rescue medication for seizure control. — Children from home group assigned to receive treatment with intranasal midazolam with doses of 0.2 mg/kg (maximum, 10 mg) body weight of the standard IV formulation of midazolam (5mg/mL) via a metered dose sprayer at 0.1 mL/spray (i.e. 0.5 mg/spray). If the volume to be administered exceeded 1 mL, the dose was divided between both nostrils to avoid runoff and swallowing
  Arms: Nasal administration of midazolam in home group
Drug: administration of Buccal midazolam in home group as a rescue medication for seizure control. — Children from home group randomly assigned to receive treatment with buccal midazolam with doses of 0.2 mg/kg (maximum, 10 mg) body weight of the standard IV formulation of midazolam (5mg/mL) via dripping between the cheek and the gum per side using insulin syringe
  Arms: buccal administration of midazolam in home group
Drug: administration of intramuscular midazolam in homegroup as a rescue medication for seizure control. — Children from home group randomly assigned to receive treatment with intramuscular midazolam with doses of 0.2 mg/kg (maximum, 10 mg) body weight of the standard IV formulation of midazolam (5mg/mL) using 3 mm syringe in the front aspect of thigh
  Arms: intramuscular administration of midazolam in home group
Drug: administration of Nasal midazolam in ER group as a rescue medication for seizure control. — Children from the ER group assigned to receive treatment with intranasal midazolam with doses of 0.2 mg/kg (maximum, 10 mg) body weight of the standard IV formulation of midazolam (5mg/mL) via a metered dose sprayer at 0.1 mL/spray (i.e. 0.5 mg/spray). If the volume to be administered exceeded 1 mL, the dose was divided between both nostrils to avoid runoff and swallowing
  Arms: Nasal administration of midazolam in ER group
Drug: administration of Buccal midazolam in ER group as a rescue medication for seizure control. — Children from ER group randomly assigned to receive treatment with buccal midazolam with doses of 0.2 mg/kg (maximum, 10 mg) body weight of the standard IV formulation of midazolam (5mg/mL) via dripping between the cheek and the gum per side using insulin syringe
  Arms: buccal administration of midazolam in ER group
Drug: administration of intramuscular midazolam in ER group as a rescue medication for seizure control. — Children from ER group randomly assigned to receive treatment with intramuscular midazolam with doses of 0.2 mg/kg (maximum, 10 mg) body weight of the standard IV formulation of midazolam (5mg/mL) using 3 mm syringe in the front aspect of thigh
  Arms: Intramuscular administration of midazolam in ER group

SUMMARY:
A randomized controlled clinical trial comparing patient/ ER physician satisfaction and ease of administration of 3 non IV routes of midazolam as a rescue medication for seizure control. Study population included children with known seizure disorder who were prescribed midazolam by pediatric neurologist at home and those presenting to ER with following inclusion and exclusion criteria

DETAILED DESCRIPTION:
Recruited patients randomized using previously computer-generated randomization tables prepared by expert statistician. Study was approved by the faculty ethical committee prior to its start and oral informed consent was obtained from the parents. In order to simplify the administration process a reference guide was prepared for doses according to weight for each of the 3 routes.

Two major groups were included (home and ER group) and each were subdivided into 3 groups according to route of administration

Children was randomly assigned to receive treatment with intranasal, intramuscular or buccal midazolam with doses of 0.2 mg/kg (maximum, 10 mg) body weight of the standard IV formulation of midazolam (5mg/mL) .Intranasal form was administered via a metered dose sprayer at 0.1 mL/spray (i.e. 0.5mg/spray). If the volume to be administered exceeded 1 mL, then the dose was divided between both nostrils to avoid runoff and swallowing. Administration was via sprays in each nostril (for nasal) or dripping between the cheek and the gum per side using insulin syringe (for buccal) or using 3 mm syringe in the front aspect of thigh for intramuscular injection.

Caretakers who gave the study medication recorded their observations and answered a series of questions regarding time to drug administration, seizure cessation time, seizure recurrence, need for hospitalization or ER visits and any encountered difficulties or side effects. Ease of administration of was rated using a scale prepared by expert statistian from very easy to very difficult and overall satisfaction with the medication was rated using 10-point nominal scale (0, being not satisfied and 10, greatly satisfied). Seizures that did not cease for ten minutes after drug administration and the need to use additional medication was categorized as a treatment failure criteria.

Recruited caretakers who did not spontaneously report the use of the study medication were contacted by phone monthly to address any questions and to remind them of the study. Problems with different routes of delivery were discussed, for example excessive head movements, ryle or upper respiratory tract infections and where possible suggestions and advices to help with addressed issue was provided .If a caretaker reported use of study medication at the time of the phone call, information was obtained at that time. In this group, not all children received a benzodiazepine because of different reasons: unavailability of the drug at home or at school, spontaneous resolution of seizures, difficulty in administrating the drug, or panic.

ER doctor given a brief survey after the administration to evaluate sedation, discomfort and other adverse effects of the medication as well as any administration difficulties and data for other secondary outcomes (need for additional medical support, hospitalization, repeated seizures…etc).

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 1 months and 17 years
* children with known seizure disorder who were prescribed midazolam by pediatric neurologist at home
* Patients with generalized tonic-clonic status epilepticus with seizures accompanied by loss of consciousness with any of the following characteristics persistent at the time of study drug administration:

  1. Currently presenting with seizure (convulsive) activity and 3 or more convulsions within the preceding hour
  2. Currently presenting with seizure (convulsive) and 2 or more convulsions in succession without recovery of consciousness
  3. Currently presenting with a single seizure (convulsive) lasting >=5 minutes

Exclusion Criteria:

* Any child who had received an anticonvulsant benzodiazepine agent within 1 hour of presentation
* Patients with known history of hypersensitivities, non-responsiveness or contraindications to benzodiazepines (i.e., clinically significant respiratory depression, severe acute hepatic failure, myasthenia gravis, syndrome of sleep apnea, glaucoma with closed angle, use of concomitant drugs determined by the investigator to have a contraindication to the use of bbenzodiazepines.)
* Patients with significant hypotension and cardiac dysrhythmia (e.g. atrioventricular block of second or third degree, ventricular tachycardia]).
* Patients with current hypoglycemia (glucose <60 milligram per deciliter [mg/dl]) on presentation at the hospital or healthcare setting.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 305 (Actual)
Dates: Start 2019-01-19 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with therapeutic success | 30 minutes post drug administration
  Percentage of participants with therapeutic success defined as cessation of visible seizure activity within 10 minutes (mins) with a sustained absence of visible seizure activity for 30 minutes following a single dose of anticonvulsant agent time frame: from start drug administration up to 30 minutes postdose ] i.e Successful responder (onset of seizure cessation within 10 minutes or duration of seizure control >30 minutes without seizure relapse), or Unsuccessful/nonresponder (onset of seizure cessation >10 minutes or duration of seizure control <30 minutes

SECONDARY OUTCOMES:
sustained absence of seizure activity for at least 1 hour | from start of study drug administration up to 1 hour postdose
  Percentage of participants whose seizure event stopped within 10 minutes of single dose of anticonvulsant and who have sustained absence of seizure activity for at least 1 hour
sustained absence of seizure activity for 4 hour | from start of study drug administration up to 4 hours postdose
  Percentage of participants whose seizure event stopped within 10 minutes of single dose of anticonvulsant and who have sustained absence of seizure activity for at least 4 hours
sustained absence of seizure activity for 6 hour | from start of study drug administration up to 6 hours postdose
  Percentage of participants whose seizure event stopped within 10 minutes of single dose of anticonvulsant and who have sustained absence of seizure activity for at least 6 hours
Time to resolution of seizures (convulsions) | 30 minutes
  Time to resolution of seizures (convulsions) after drug administration Cessation of seizure activity was defined as caregiver/physician-confirmed cessation of abnormal motor activity with at least partial recovery of consciousness
Time of drug preparation and administration | 45 minutes
  time taken to prepare and administer drug
Emergency department visits | 24 hours post drug administration
  Number of patients from home group who needed to go to ER after drug adminstration
percentage of patients admitted to hospital | 24 hours post drug administration
  Number of patients that were admitted to the hospital or intensive care unit after their seizure and use of study medication.
need for additional doses or additional drugs for seizure control | 10 minutes post drug administration
  Percentage of participants who required additional anticonvulsant medication for ongoing status epilepticus (se) 10 minutes after single dose administration of anticonvulsant
Seizure recurrence at 1 ,4 , 6 and 24 hrs | 24 hours post drug administration
  Seizure recurrence at 1 ,4 , 6 and 24 hrs of cessation of presenting convulsion
Respiratory depression | 6 hours post drug administration
  persistent decrease in oxygen saturation to <92% measured at 0, 10 minutes, 30 minutes, and 1, 4 , 6 hrs postdose (ie, <92% on room air for 2 minutes or more after dosing while monitoring aspiration pneumonia
Sedation or agitation | 4 hours post drug administration
  • Sedation or agitation measured by a 7 point nominal scale where 1 represented deep sedation and 7 sever agitation
Frequency of cardio-respiratory side effects | 6 hours post drug administration
  Frequency of cardio-respiratory side effects development of hypotension (fall of >/= 20 mmhg systolic and/ or >/= 10 mmhg diastolic pressure) within 0, 10 and 30 mins, 1, 4 , 6 hrs postdose of drug administration
Occurrence of route of administration and benzodiazepine related side effects | 6 hours post drug administration
  Adverse events, including but not limited nasal irritation, dizziness, Stuffy nose, headache , nausea, agitation , cardiopulmonary dysfunction, ataxia, and abnormal vital signs were recorded
Caretakers and physicians ease of administration and satisfaction with the medication | up to 1 months after drug administration
  Ease of administration of was rated using a scale prepared by expert statistician from very easy to very difficult and overall satisfaction with the medication was rated using 10-point nominal scale (0, being not satisfied and 10, greatly satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Omnia El Rashidy, MD, Study Chair — Ain Shams University; Iman Ali, MD, Study Chair — Ain Shams University; Maha El Gafary, MD, Study Chair — Ain Shams University; Maha zakariya Mohammed, MD, Study Chair — Ain Shams University; Rana El Garhy, master, Principal Investigator — Ministry of Health
Locations (1):
- Ain Shams Pediatric hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No